CLINICAL TRIAL: NCT05489783
Title: Glioma Developmental and HyperActive Ras Tumor (DHART) Board
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 22-199
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Glioma
Keywords: NF1-associated glioma; Neurofibromatosis; Registry; 22-199
MeSH Terms: conditions — Glioma; Neurofibromatoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will collect medical records, scan results, and complete surveys to create a registry about people with a neurofibromatosis type 1-associated brain tumor (NF1-associated glioma). A registry is a collection of health information about individuals, and it is usually focused on a specific diagnosis or condition.

This registry study will help the researchers learn more about the diagnosis, treatment, and quality of life of people with NF1-associated glioma. The researchers want to understand what happens as a result of different treatments for NF1-associated glioma and how these treatments and the disease itself affect people's lives over a period of time. Information collected during this study could affect how doctors diagnose, test, and treat NF1-associated glioma, and the study could help future patients with this type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis that meets NIH criteria for NF1 disease by either 1) documented clinical record establishing NF1 or 2) self-reported with supported documentation upon medical record collection.
* Willing to have historical and future NF1 related health records sent to registry for review.
* Radiologic or pathologically confirmed glioma.
* Individuals ≥18 years of age on the date of informed consent.

Exclusion Criteria:

* Unwillingness to sign informed consent.
* No proficiency in English or Spanish as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NF1 glioma will be enrolled in this registry study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Registry of patients with Neurofibromatosis Type 1 (NF1) associated glioma | 5 years
  The overarching goal of the registry is to collect baseline and follow-up 1) clinical and 2) imaging data to have a centralized and living repository of information about the adult glioma NF1 patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Piotrowski, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering West Harrison (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/